CLINICAL TRIAL: NCT06816810
Title: TALLman Family Energizes Research To Help Alleviate Neuroinflammation in Parkinson's Disease - "TALLER THAN PD." A Phase 2 Futility Study to Evaluate the Efficacy, Safety and Tolerability of Hydroxychloroquine in Subjects With Early Treated Parkinson's Disease
Brief Title: A Study to Evaluate Efficacy, Safety and Tolerability of Hydroxychloroquine in Subjects With Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Taller Than PD
Record Dates: First submitted 2025-01-14; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Parkinson&Amp;#39;s Disease
Keywords: Hydroxychloroquine; Neuroinflammation; Neuroprotection; Parkinson
MeSH Terms: conditions — Neuroinflammatory Diseases | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydroxychloroquine Treatment for Early Parkinson's Disease (HCQ-PD) (Experimental): This is an open-label study where 40 participants with early-treated Parkinson's Disease will be receive 200mg of Hydroxychloroquine, orally, twice daily for 48 weeks.
  Interventions: Drug: Hydroxychloroquine (HCQ)

INTERVENTIONS:
Drug: Hydroxychloroquine (HCQ) — The intervention involves hydroxychloroquine (HCQ), administered orally in 200 mg tablets, with a dosing schedule of 200 mg twice daily (400 mg per day). The treatment duration is 48 weeks, after which participants will enter a 4-week safety follow-up period. HCQ will be taken alongside stable doses of Parkinson's disease (PD) medications, with no anticipated changes during the study. Monitoring for adverse events, laboratory assessments, and efficacy evaluations will occur regularly throughout the 12-month period. The study does not include a placebo group or other treatment arms.

SUMMARY:
The purpose of this study is to determine if hydroxychloroquine is safe to take and whether there is potential for it to slow the progression of PD symptoms. This will be done by comparing how PD symptoms progress throughout the study compared to how people with PD typically progress. Within PD, it is thought that an inflammation response is associated with abnormal forms of a protein called alpha-synuclein in the brain. Individuals who have taken this medication for other conditions have been shown to be less likely to develop PD than people who have not taken this medication. Therefore, it is hoped that the study drug may interrupt the inflammation response and in turn stop/delay the progression of PD.

DETAILED DESCRIPTION:
Parkinson disease (PD) is a progressive neurodegenerative disorder pathologically characterized by the loss of dopaminergic neurons in the substantia nigra and the presence of α-synuclein protein inclusions termed Lewy bodies. There is increasing evidence of the important role of inflammation in the pathophysiology in PD. Studies of the innate and adaptive immune systems provide evidence that immune dysregulation in both the periphery and brain can cause upregulation of inflammatory cytokines that initiate a cascade of pro-inflammatory signaling events that ultimately result in the neurotoxicity. Post-mortem studies reveal activated microglia and T-cells and immunoglobulin deposition in brain tissue from PD subjects. Alterations in immune cells are detected in living PD subjects, with most consistent findings pointing to T-cell and monocyte changes. Peptides derived from αsynuclein, the key protein that aggregates in PD and the primary component of Lewy bodies, can activate T-cells from PD patients. Pro-inflammatory cytokines and chemokines are elevated in blood and cerebrospinal fluid (CSF) specimens from PD subjects. In vivo evaluation of microglial activity has been performed using positron emission tomography (PET) ligands to measure and shown evidence of neuroinflammation in the brains of patients with PD. Mutations in more than 20 genes have been identified that cause PD with many of them (e.g. LRRK2, SNCA, GBA, PRKN, PINK1) encoding proteins that modulate immune function. Animal PD models show inflammatory changes, and manipulation of inflammation can alter neurodegeneration in animal models. A wide range of epidemiologic studies have supported the role of inflammation in PD that includes data to suggest that ibuprofen and treatment of inflammatory bowel disease with anti- tumor necrosis factor (TNF) biologics are associated with reduced PD risk.

The repurposing of generic drugs is a strategy to identify new treatment options for PD because of their known safety profile. Hydroxychloroquine (HCQ) was approved for medical use for over 50 years as a treatment for malaria, systemic lupus erythematosus, and rheumatoid arthritis and is on the World Health Organization's List of Essential Medicines. It belongs to a class of medications known as disease-modifying antirheumatic drug that can reduce skin problems in lupus and prevent swelling/pain in arthritis. It has been shown to interfere with lysosomal activity and autophagy, interact with membrane stability and alter signaling pathways and transcriptional activity, which can result in inhibition of cytokine production and modulation of certain co-stimulatory molecules. HCQ has been studied in multiple sclerosis (MS) which is an inflammatory and neurodegenerative disease of the central nervous. In mice models of MS, HCQ has been shown to inhibit microglia activation and attenuate the severity of disease. Hydroxychloroquine reduces microglial activity and attenuates experimental autoimmune encephalomyelitis. A phase II futility trial of 200 mg bid HCQ in 35 patients with primary progressive MS was associated with reduced disability worsening over 18 months. HCQ was well tolerated overall, with adverse events in 82% and serious adverse events in 12% of participants. All serious adverse events were felt to be unlikely related to HCQ. In this study, HCQ treatment attenuated the increase of neurofilament-light (NfL) after 6 months of treatment and up to 18 months of follow-up, suggesting a treatment effect of HCQ over these biomarkers

ELIGIBILITY:
Inclusion Criteria:

* The subject is ≥35 and ≤80 years of age at the time of informed consent.
* The subject has a clinical diagnosis of PD for at least 6 months and for no longer than 4 years before initiation of screening as confirmed by a neurologist using the MDS Criteria for Parkinson's Disease (Postuma, Berg et al. 2015)
* The subject has a Hoehn and Yahr score ≤2.
* The subject has been on stable doses of PD medications for at least 30 days and the investigator does not anticipate they will require a change of their usual PD medications for a period of 48 weeks.
* The subject has a score ≥24 on the MoCA scale.
* The subject does not have severe motor fluctuations or disabling dyskinesias in the clinical judgment of the investigator (MDS-UPDRS score > 2 on any item IV).
* If a sexually active man or a woman of childbearing potential, the subject agrees to use highly effective birth control or to remain abstinent during the trial and for 30 days after the last dose of HCQ. Acceptable (highly effective) methods of contraception for this study include hormonal contraceptives or implant); intrauterine device or system; complete abstinence from sexual intercourse if this is the subject's usual and preferred lifestyle; or sexual partner with surgical sterilization (e.g., tubal ligation, hysterectomy and/or bilateral oophorectomy, vasectomy).
* The subject is capable of giving signed informed consent, which includes understanding the purpose and risks of the study, compliance with the requirements and restrictions that are listed in the informed consent form (ICF) and this protocol, and authorization to use confidential health information in accordance with national and local subject privacy regulations

Exclusion Criteria:

* The subject has atypical or secondary parkinsonism by medical history or in the opinion of the investigator. Atypical parkinsonism includes, but is not limited to, diagnoses of progressive supranuclear palsy, cortico-basal syndrome, and multiple system atrophy. Secondary parkinsonism includes drug-induced, toxin-induced, postinfectious, posttraumatic, or vascular parkinsonism.
* The subject has a history of (within 60 days before initiation of screening) or has planned upcoming major surgery that could interfere with, or for which the treatment might interfere with, the conduct of the study or that would pose an unacceptable risk to the subject in the opinion of the investigator.
* The subject has any active or chronic disease including but not limited to cardiomyopathy or condition other than PD that could interfere with, or for which the treatment might interfere with, the conduct of the study or pose an unacceptable risk to the subject in the opinion of the investigator based on medical history, physical examination, vital signs, 12-lead ECG, or clinical laboratory tests.
* Minor deviations of laboratory values from the normal range may be acceptable if judged by the investigator to have no/minor clinical relevance.
* The subject has a recent history (last 6 months) of abuse of addictive substances (alcohol, illegal substances), currently uses >21 units of alcohol per week, or is a regular recreational user of sedatives, hypnotics, tranquillizers, or any other addictive agent in the opinion of the investigator.
* The subject is currently pregnant, is planning pregnancy within the timeframe of the study, or is breastfeeding.
* Patient has a history of psoriasis or porphyria.
* The subject has used any of the following medications within 60 days before Baseline: typical or atypical antipsychotics (including, but not limited to, clozapine, pimavanserin, olanzapine, risperidone, and aripiprazole), metoclopramide, prochlorperazine, methyldopa, tetrabenazine, azithromycin, antimalarial drugs, tamoxifen, amiodarone, dapsone, or digoxin.
* The subject has received a vaccination within 14 days before administration of the first dose of IMP.
* The subject has a prior history of or there is a plan to undergo Deep Brain stimulation, brain lesional procedures (i.e., thalamotomy), or focused ultrasound; to initiate gene therapy treatment for PD; or to initiate use of any formulation of intestinal infusion or continuous subcutaneous infusion of PD medications during the following 48 weeks.
* The subject is currently participating in or has participated in an investigational drug study within 3 months or 5 half-lives, whichever is longer; in a therapeutic device study within 3 months before the first dose of IMP; or has previously participated in a gene therapy trial. Concurrent participation in an observational study is acceptable.
* The subject has renal insufficiency as defined by an estimated glomerular filtration rate (eGFR) of <60 mL/min at screening.
* The subject has cirrhosis or any of the following laboratory values at screening: serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 times the upper limit of normal (ULN) or bilirubin >2 × ULN except if the subject has known or suspected Gilbert's disease.
* The subject has a QTcF (QT interval corrected for heart rate by Fridericia's method) value >450 msec if male or >470 msec if female at screening.
* The subject has previously received hydroxychloroquine or has a known allergy or hypersensitivity to hydroxychloroquine or any components of the formulation.
* The subject has a history of bone marrow failure, anemia, aplastic anemia, agranulocytosis, leukopenia, or thrombocytopenia
* The subject has a history of glucose-6-phosphate dehydrogenase (G-6-PD) deficiency
* The subject is unable or unlikely to comply with the dosing schedule or study evaluations in the judgment of the investigator.
* The subject is a member of a protected/vulnerable population, defined as persons who are pregnant, parturient, or breastfeeding; persons who are deprived of liberty; persons who are admitted to a health or social institution for purposes other than research; adults who are under legal protection or who are unable to express their consent; persons who are in an emergency situation and are unable to express their prior consent; and persons are who are non-affiliated or a non-beneficiary of a social security system.
* The subject is a relative of the investigator or sponsor or the relative of an employee of the sponsor.
* The subject has a history of retinopathy or is found to have a significant retina finding on screening ophthalmologic examination.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Throughout enrollment (4 weeks of screening) to the end of treatment at 48 weeks and 4-week safety follow-up.
  All participants exposed to HCQ at least once will be assessed for:
  * Incidence and severity of treatment-emergent adverse events (TEAEs)
  * Relationship of TEAEs to HCQ
  * Percentage of discontinuations due to adverse events (AEs)
Efficacy of Hydroxychloroquine (HCQ) in Delaying Clinical Motor Progression Using MDS-UPDRS Part III | Throughout enrollment to the end of treatment at 48 weeks. MDS-UPDRS Part III will be evaluated at baseline, 24 weeks and 48 weeks.
  Another primary clinical outcome is assess change in motor symptom severity, specifically using the movement disorder society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III. A ≥4-point increase (one standard deviation) over 48 weeks will be used as a threshold to assess whether HCQ delays clinical motor progression of PD when compared to historical controls.

SECONDARY OUTCOMES:
Efficacy of Hydroxychloroquine (HCQ) in Delaying Clinical PD Progression Using CGI-C Scale | Throughout enrollment to the end of treatment at 48 weeks. CGI-C will be evaluated at baseline, 24 weeks and 48 weeks.
  The Clinical Global Impression of Change (CGI-C) scale assesses the clinician's perception of the change in a patient's condition. It ranges from 1 (very much improved) to 7 (very much worse). A score of 1-3 indicates improvement, while a score of 5-7 indicates worsening of the condition. This study will identify the number of participants with worsening CGI-C scale by the end of the study.
Efficacy of Hydroxychloroquine (HCQ) in Delaying Clinical PD Progression Using CGI-S Scale | Throughout enrollment to the end of treatment at 48 weeks. CGI-S will be evaluated at baseline, 24 weeks and 48 weeks.
  The Clinical Global Impression-Severity (CGI-S) scale will be used to assess the severity of Parkinson's disease symptoms based on clinician judgment. The scale ranges from 1 (normal, not at all ill) to 7 (extremely ill). A higher score indicates more severe symptoms. A reduction in score will indicate an improvement in disease severity. This study will identify the number of participants with worsening CGI-S scale by the end of the study.
Efficacy of Hydroxychloroquine (HCQ) in Delaying Clinical PD Progression Using PGI-S Scale | Throughout enrollment to the end of treatment at 48 weeks. PGI-S will be evaluated at baseline, 24 weeks and 48 weeks.
  The Patient Global Impression-Severity (PGI-S) scale measures the patient's assessment of the severity of their Parkinson's disease symptoms at the time of the assessment. The scale ranges from 1 (not at all ill) to 7 (extremely ill). A higher score indicates greater severity, and a decrease in score over time indicates improvement. This study will identify the number of participants with worsening PGI-S scale by the end of the study.
Efficacy of Hydroxychloroquine (HCQ) in Delaying Clinical PD Progression Using PGI-C Scale | Throughout enrollment to the end of treatment at 48 weeks. PGI-C will be evaluated at baseline, 24 weeks and 48 weeks.
  The Patient Global Impression of Change (PGI-C) measures the patient's own perception of how much their condition has changed since the beginning of the study. The scale ranges from 1 (very much improved) to 7 (very much worse), with 1-3 indicating improvement and 5-7 indicating worsening. This study will identify the number of participants with worsening PGI-C scale by the end of the study.
Change in Quality of Life (QoL) as assessed by the PDQ-8 | Throughout enrollment to the end of treatment at 48 weeks. QoL will be evaluated at baseline, 24 weeks and 48 weeks.
  The Parkinson's Disease Questionnaire-8 (PDQ-8) will be used to assess changes in quality of life (QoL) over the 48-week treatment period. The PDQ-8 is a shorter version of the PDQ-39 and includes 8 items measuring physical functioning, emotional well-being, and social participation. Scores range from 0 to 32, where a higher score indicates worse quality of life. A decrease in the score reflects an improvement in QoL.
Efficacy of Hydroxychloroquine (HCQ) Using Change in Modified Hoehn and Yahr Scale | Throughout enrollment to the end of treatment at 48 weeks. Modified Hoehn and Yahr Scale will be evaluated at baseline, 24 weeks and 48 weeks.
  The Modified Hoehn and Yahr Scale is widely recognized for tracking the progression of Parkinson's disease and is crucial for evaluating treatment effects on motor symptoms. It will measure disease severity in Parkinson's patients, ranging from 0 (no signs of disease) to 5 (wheelchair-bound or bedridden unless aided). A decrease in score indicates an improvement in motor function and disease severity.
Efficacy of Hydroxychloroquine (HCQ) in Slowing Clinical Disease Progression as Assessed by the MDS-UPDRS | Throughout enrollment to the end of treatment at 48 weeks. MDS-UPDRS will be evaluated at baseline, 24 weeks and 48 weeks.
  Movement Disorder Society-Unified Parkinson's Disease Rating Scale ( MDS-UPDRS) is a comprehensive scale for assessing both motor and non-motor aspects of Parkinson's disease. The efficacy of HCQ in slowing clinical disease progression will be measured by the change from baseline to Week 48 in various MDS-UPDRS sub-scales:
  MDS-UPDRS Part I score (Non-motor aspects of PD) MDS-UPDRS Part II score (Motor experiences of daily living) MDS-UPDRS Part III score (Motor examination) MDS-UPDRS Part II + Part III (Tremor items) MDS-UPDRS Part II + Part III (Non-Tremor items)

OTHER OUTCOMES:
Change in Motor Score as Assessed by the PRIMS Digital Assessment | Throughout enrollment to the end of treatment at 48 weeks. PRIMS Digital Assessment will be evaluated at baseline, 24 weeks and 48 weeks.
  Time from baseline to clinically meaningful progression on motor signs of the disease, as assessed by a >= 4 point increase in the MDS-UPDRS part III score (one standard deviation) in comparison to historical controls.
Change in Motor Function as Assessed by Celestra Gait Assessment | Throughout enrollment to the end of treatment at 48 weeks. Celestra insole gait assessment will be evaluated at baseline, 24 weeks and 48 weeks.
  * Adherence: Measured by analyzing the total number of tasks completed, divided by the total number of tasks prompted
  * Percent change from baseline of gait metrics/composite score generated from gait measures using Celestra insole sensors

CONTACTS AND LOCATIONS:
Overall Officials: David Grimes, MD, FRCPC, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Galna B, Lord S, Burn DJ, Rochester L. Progression of gait dysfunction in incident Parkinson's disease: impact of medication and phenotype. Mov Disord. 2015 Mar;30(3):359-67. doi: 10.1002/mds.26110. Epub 2014 Dec 27. PMID 25546558
- [Background] Gisondi P, Piaserico S, Bordin C, Bellinato F, Tozzi F, Alaibac M, Girolomoni G, Naldi L. The safety profile of hydroxychloroquine: major cutaneous and extracutaneous adverse events. Clin Exp Rheumatol. 2021 Sep-Oct;39(5):1099-1107. doi: 10.55563/clinexprheumatol/styx9u. Epub 2021 Feb 15. PMID 33635229
- [Background] Harms AS, Ferreira SA, Romero-Ramos M. Periphery and brain, innate and adaptive immunity in Parkinson's disease. Acta Neuropathol. 2021 Apr;141(4):527-545. doi: 10.1007/s00401-021-02268-5. Epub 2021 Feb 8. PMID 33555429
- [Background] Hedya SA, Safar MM, Bahgat AK. Hydroxychloroquine antiparkinsonian potential: Nurr1 modulation versus autophagy inhibition. Behav Brain Res. 2019 Jun 3;365:82-88. doi: 10.1016/j.bbr.2019.02.033. Epub 2019 Feb 22. PMID 30797853
- [Background] Holden SK, Finseth T, Sillau SH, Berman BD. Progression of MDS-UPDRS Scores Over Five Years in De Novo Parkinson Disease from the Parkinson's Progression Markers Initiative Cohort. Mov Disord Clin Pract. 2018 Jan-Feb;5(1):47-53. doi: 10.1002/mdc3.12553. Epub 2017 Sep 22. PMID 29662921
- [Background] Hooks M, Bart B, Vardeny O, Westanmo A, Adabag S. Effects of hydroxychloroquine treatment on QT interval. Heart Rhythm. 2020 Nov;17(11):1930-1935. doi: 10.1016/j.hrthm.2020.06.029. Epub 2020 Jun 28. PMID 32610165
- [Background] Huang L, Li Q, Shah SZA, Nasb M, Ali I, Chen B, Xie L, Chen H. Efficacy and safety of ultra-short wave diathermy on COVID-19 pneumonia: a pioneering study. Front Med (Lausanne). 2023 Jun 5;10:1149250. doi: 10.3389/fmed.2023.1149250. eCollection 2023. PMID 37342496
- [Background] Imanova Yaghji N, Kan EK, Akcan S, Colak R, Atmaca A. Hydroxychloroquine Sulfate Related Hypoglycemia In A Non-Diabetic COVID-19 Patient: A Case Report and Literature Review. Postgrad Med. 2021 Jun;133(5):548-551. doi: 10.1080/00325481.2021.1889820. Epub 2021 Feb 26. PMID 33583332
- [Background] Jarzyna R, Kiersztan A, Lisowa O, Bryla J. The inhibition of gluconeogenesis by chloroquine contributes to its hypoglycaemic action. Eur J Pharmacol. 2001 Oct 12;428(3):381-8. doi: 10.1016/s0014-2999(01)01221-3. PMID 11689198
- [Background] Kwak YT, Yang Y, Park SY. Chloroquine-associated psychosis mimicking very late-onset schizophrenia: Case Report. Geriatr Gerontol Int. 2015 Aug;15(8):1096-7. doi: 10.1111/ggi.12490. No abstract available. PMID 26391537
- [Background] Li D, Hong X, Chen T. Association Between Rheumatoid Arthritis and Risk of Parkinson's Disease: A Meta-Analysis and Systematic Review. Front Neurol. 2022 May 11;13:885179. doi: 10.3389/fneur.2022.885179. eCollection 2022. PMID 35645965
- [Background] Lipner SR, Wang Y. Retrospective analysis of dermatologic adverse events associated with hydroxychloroquine reported to the US Food and Drug Administration. J Am Acad Dermatol. 2020 Nov;83(5):1527-1529. doi: 10.1016/j.jaad.2020.07.007. Epub 2020 Jul 8. No abstract available. PMID 32652194
- [Background] Liu SY, Qiao HW, Song TB, Liu XL, Yao YX, Zhao CS, Barret O, Xu SL, Cai YN, Tamagnan GD, Sossi V, Lu J, Chan P. Brain microglia activation and peripheral adaptive immunity in Parkinson's disease: a multimodal PET study. J Neuroinflammation. 2022 Aug 29;19(1):209. doi: 10.1186/s12974-022-02574-z. PMID 36038917
- [Background] Murray JJ, Lee MS. Re: Marmor et al.: American Academy of Ophthalmology Statement: Recommendations on screening for chloroquine and hydroxychloroquine retinopathy (2016 Revision). (Ophthalmology 2016;123:1386-1394). Ophthalmology. 2017 Mar;124(3):e28-e29. doi: 10.1016/j.ophtha.2016.06.062. No abstract available. PMID 28219513
- [Background] McGhie TK, Harvey P, Su J, Anderson N, Tomlinson G, Touma Z. Electrocardiogram abnormalities related to anti-malarials in systemic lupus erythematosus. Clin Exp Rheumatol. 2018 Jul-Aug;36(4):545-551. Epub 2018 Apr 13. PMID 29652656
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] O'Laughlin JP, Mehta PH, Wong BC. Life Threatening Severe QTc Prolongation in Patient with Systemic Lupus Erythematosus due to Hydroxychloroquine. Case Rep Cardiol. 2016;2016:4626279. doi: 10.1155/2016/4626279. Epub 2016 Jul 12. PMID 27478650
- [Background] Paakinaho A, Koponen M, Tiihonen M, Kauppi M, Hartikainen S, Tolppanen AM. Disease-Modifying Antirheumatic Drugs and Risk of Parkinson Disease: Nested Case-Control Study of People With Rheumatoid Arthritis. Neurology. 2022 Mar 22;98(12):e1273-e1281. doi: 10.1212/WNL.0000000000013303. Epub 2022 Jan 21. PMID 35064025
- [Background] Peter I, Dubinsky M, Bressman S, Park A, Lu C, Chen N, Wang A. Anti-Tumor Necrosis Factor Therapy and Incidence of Parkinson Disease Among Patients With Inflammatory Bowel Disease. JAMA Neurol. 2018 Aug 1;75(8):939-946. doi: 10.1001/jamaneurol.2018.0605. PMID 29710331
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Qin H, Buckley JA, Li X, Liu Y, Fox TH 3rd, Meares GP, Yu H, Yan Z, Harms AS, Li Y, Standaert DG, Benveniste EN. Inhibition of the JAK/STAT Pathway Protects Against alpha-Synuclein-Induced Neuroinflammation and Dopaminergic Neurodegeneration. J Neurosci. 2016 May 4;36(18):5144-59. doi: 10.1523/JNEUROSCI.4658-15.2016. PMID 27147665
- [Background] Samii A, Etminan M, Wiens MO, Jafari S. NSAID use and the risk of Parkinson's disease: systematic review and meta-analysis of observational studies. Drugs Aging. 2009;26(9):769-79. doi: 10.2165/11316780-000000000-00000. PMID 19728750
- [Background] Schrezenmeier E, Dorner T. Mechanisms of action of hydroxychloroquine and chloroquine: implications for rheumatology. Nat Rev Rheumatol. 2020 Mar;16(3):155-166. doi: 10.1038/s41584-020-0372-x. Epub 2020 Feb 7. PMID 32034323
- [Background] Spillantini MG, Schmidt ML, Lee VM, Trojanowski JQ, Jakes R, Goedert M. Alpha-synuclein in Lewy bodies. Nature. 1997 Aug 28;388(6645):839-40. doi: 10.1038/42166. No abstract available. PMID 9278044
- [Background] Srinivasa A, Tosounidou S, Gordon C. Increased Incidence of Gastrointestinal Side Effects in Patients Taking Hydroxychloroquine: A Brand-related Issue? J Rheumatol. 2017 Mar;44(3):398. doi: 10.3899/jrheum.161063. No abstract available. PMID 28250164
- [Background] Sterling NW, Cusumano JP, Shaham N, Piazza SJ, Liu G, Kong L, Du G, Lewis MM, Huang X. Dopaminergic modulation of arm swing during gait among Parkinson's disease patients. J Parkinsons Dis. 2015;5(1):141-50. doi: 10.3233/JPD-140447. PMID 25502948
- [Background] Wilson J, Alcock L, Yarnall AJ, Lord S, Lawson RA, Morris R, Taylor JP, Burn DJ, Rochester L, Galna B. Gait Progression Over 6 Years in Parkinson's Disease: Effects of Age, Medication, and Pathology. Front Aging Neurosci. 2020 Oct 15;12:577435. doi: 10.3389/fnagi.2020.577435. eCollection 2020. PMID 33192470
- [Background] Yacoubian TA, Fang YD, Gerstenecker A, Amara A, Stover N, Ruffrage L, Collette C, Kennedy R, Zhang Y, Hong H, Qin H, McConathy J, Benveniste EN, Standaert DG. Brain and Systemic Inflammation in De Novo Parkinson's Disease. Mov Disord. 2023 May;38(5):743-754. doi: 10.1002/mds.29363. Epub 2023 Feb 28. PMID 36853618